CLINICAL TRIAL: NCT05715957
Title: Influence of X- Chromosome Activation Pattern in Muscles on Symptoms and Progression of Cardiac and Muscle Symptoms Signs in Women With Pathogenic Dystrophin Gene Variants: A 6-year Follow-up of 53 Patients
Brief Title: Follow-up Study on Female Carriers With DMD Gene Variants
Status: Enrolling by invitation | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Zhe Lyu, MD,PhD student, Rigshospitalet, Denmark
Other Study IDs: 98434
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Muscular Dystrophy; Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: XCI; follow up; MRI; spectroscopy
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests:
  Blood samples will be drawn and analyzed for cardiac markers (myoglobin, creatine kinase, creatine kinase MB, pro-brain natriuretic peptide (proBNP), and troponin T (TnT)) and proteomics.
  Biopsy procedure:
  Muscle biopsies will be sent to the Department of Clinical Genetics (Rigshospitalet) for genetic analysis to investigate the X-chromosome inactivation pattern. No other genetic information will be obtained during these tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- female carriers of DMD gene variants
  Interventions: Other: No intervention
- patients with BMD
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background Duchenne and Becker muscular dystrophies are X-linked recessive allelic disorders caused by mutations of the dystrophin gene on chromosome Xp21. Female carriers may pass on the pathogenic variant to their daughters, resulting in a significant number of female carriers of pathogenic DMD variants. There was a large variability in the severity of symptoms with some being asymptomatic and some having severe symptoms. Skewed X-Chromosome Inactivation (XCI) might explain some of this variability. But now, the underlying cause of the large variability in phenotype is therefore uncertain.

Aim

1. To describe the change over a 6-year follow-up period in the structure and function of the heart and in function and muscle fat fraction in skeletal muscle of DMD/BMD carriers.
2. To explain the relationship between the XCI and the severity of the disease (phenotype).
3. To compare cardiac affection of female carriers of DMD/BMD to patients with BMD using new cardiac MRI techniques (spectroscopy and Dixon sequences).

Methods

This study contains three parts:

Part 1 is a 6-year follow-up on 53 genetically verified female carriers of pathogenic DMD variants initially investigated in 2016-2018 at Copenhagen Neuromuscular Center, Rigshospitalet (Ethical journal no. H-16035677). In this part, the same 53 females will be investigated with the same measurements as 6 years ago to describe the progression of symptoms. All the follow-up results from this study will be compared to the results from 6 years ago.

In Part 2 a muscle biopsy will be taken from 1-3 muscles (see "3.3.3 Description of outcomes) to investigate the XCI. To correlate the XCI to the phenotype, these patients will also undergo a muscle MRI and a Medical Research Council scale score for muscle strength (MRC).

In Part 3 The cardiac structure and function in patients with BMD will be investigated using a cardiac MRI to compare the findings with that of female carriers. An MRC will carried out to investigate if the heart affection correlates to the muscle affection.

Female carriers can decide whether to participate in Part 1, Part 2, or both. Patient with BMD can only participate in Part 3.

DETAILED DESCRIPTION:
Duchenne and Becker muscular dystrophies are X-linked recessive allelic disorders caused by mutations of the dystrophin gene on chromosome Xp21. The gene mutation causes the absence or very severe reduction of dystrophin protein in the muscle cells, triggering chronic myofiber damage, inflammation, and loss of muscle fibers. Muscle tissue is replaced by fibrous and adipose tissue which further leads to necrosis, progressive muscle weakness, and loss of independent ambulation [1].

Duchenne muscular dystrophy (DMD) is one of the commonest inherited disorders of muscle. Based on a systematic review of worldwide population-based studies the pooled prevalence of DMD and BMD was 4.78 (95% CI 1.94-11.81) and 1.53 (95% CI 0.26-8.94) per 100,000 males respectively [2].

The disorders preferentially affect males due to the X-linked inheritance. Female carriers may pass on the pathogenic variant to their daughters, resulting in a significant number of female carriers of pathogenic DMD variants. A third of all new cases are caused by de novo pathogenic variants [3].

Even though female carriers have one healthy X-chromosome, they are not necessarily asymptomatic as both muscular and cardiac involvement has been reported in carriers [4-12]. These females are classified as "manifesting carriers" [13,14]. The incidence of skeletal muscle involvement among female carriers of DMD was 2.5%-19%, and of dilated cardiomyopathy (DCM) 7.3%-16.7% for DMD carriers and 0%-13.3% for BMD carriers [2], but in one of the latest cross-sectional studies with some of the most sensitive outcome measures to date 81 % showed muscle affection [4] and 62 % cardiac dysfunction [15]. Since then, cardiac MRI techniques have been further developed, why the numbers might be even higher. Patients with BMD have not even been investigated with these techniques. Cardiomyopathy in female DMD and BMD carriers can be clinically significant. Therefore, adult unaffected dystrophinopathy carriers are recommended to undergo echocardiography every 5 years according to the clinical guidelines in Europe and the United States [16,17]. Carriers with cardiac affection are often examined even more frequently. However, no one has yet investigated the rate of progression, which can make it difficult to determine the frequency of clinical visits.

In the above-mentioned studies, there was a large variability in the severity of symptoms with some being asymptomatic and some having severe symptoms. Skewed X-Chromosome Inactivation (XCI) might explain some of this variability. When the X chromosome carrying the normal DMD gene is preferentially inactivated this will in theory lead to moderate-severe muscle involvement.

Some studies have observed that DMD carriers with moderate/severe muscle involvement, exhibit a moderate or extremely skewed XCI, in particular, if presenting with an early onset of symptoms, while DMD carriers with mild muscle involvement present a random XCI [4, 18]. However, former studies have generally had a low power, investigated the XCI in blood and not muscle, and have often not investigated asymptomatic vs symptomatic patients. Some studies are inconclusive and some even contradictory and therefore no conclusions can be made [18]. Thus, the underlying cause of the large variability in phenotype is therefore uncertain.

2.2 Aim

The aims of this study are thus:

1. To describe the change over a 6-year follow-up period in the structure and function of the heart and in function and muscle fat fraction in skeletal muscle of DMD/BMD carriers.
2. To explain the relationship between the XCI and the severity of the disease (phenotype).
3. To compare cardiac affection of female carriers of DMD/BMD to patients with BMD using new cardiac MRI techniques (spectroscopy and Dixon sequences).

3. Methods 3.1 Study methods

This study contains three parts:

Part 1 is a 6-year follow-up on 53 genetically verified female carriers of pathogenic DMD variants initially investigated in 2016-2018 at Copenhagen Neuromuscular Center, Rigshospitalet (Ethical journal no. H-16035677). In this part, the same 53 females will be investigated with the same measurements as 6 years ago to describe the progression of symptoms. All the follow-up results from this study will be compared to the results from 6 years ago.

In Part 2 a muscle biopsy will be taken from 1-3 muscles (see "3.3.3 Description of outcomes) to investigate the XCI. To correlate the XCI to the phenotype, these patients will also undergo a muscle MRI and a Medical Research Council scale score for muscle strength (MRC).

In Part 3 The cardiac structure and function in patients with BMD will be investigated using a cardiac MRI to compare the findings with that of female carriers. An MRC will carried out to investigate if the heart affection correlates to the muscle affection.

Female carriers can decide whether to participate in Part 1, Part 2, or both. Patient with BMD can only participate in Part 3.

ELIGIBILITY:
Part 1:

Criteria of inclusion:

* Female gender
* Verified carrier of DMD gene mutations through genetic testing.
* Age of 18 years or more
* Participation in the study 6 years ago

Criteria of exclusion from MRI:

* Contraindications to MRI (pacemaker or other internal metal or magnetic devices)
* Claustrophobia.
* Pregnant or nursing women.
* Competing disorders and other muscle disorders, which may alter measurements of i.e., muscle strength. The investigator will decide whether or not the competing disorder can significantly influence the results.

Patients will be investigated with all other measurements than MRI if not eligible for MRI.

Part 2:

Criteria of inclusion:

* Female gender
* Verified carrier of DMD gene mutations through genetic testing.
* Age of 18 years or more

Criteria of exclusion:

• Anticoagulating medicine that cannot be paused due to health reasons

Part 3:

Criteria of inclusion:

* Genetically verified patient with BMD
* Age of 18 years or more

Criteria of exclusion:

* Contraindications to MRI (pacemaker or other internal metal or magnetic devices)
* Claustrophobia.
* Atrial fibrillation
* Competing disorders and other muscle disorders, which may alter measurements of i.e., muscle strength. The investigator will decide whether or not the competing disorder can significantly influence the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are identified from the Department of Clinical Genetics and Copenhagen Neuromuscular Center, Rigshospitalet. We aim at including the 53 carriers of DMD variants that we investigated 6 years ago for Part 1. These patients will be asked to participate in Part 2 as well (optional). If we cannot recruit 20 patients for Part 2 from Part 1 (see Power Calculation), we will recruit new patients identified from the Department of Clinical Genetics or Copenhagen Neuromuscular Center, Rigshospitalet. We need 32 patients with BMD for Part 3 (see Power Calculation), which will be recruited from Copenhagen Neuromuscular Center, Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in fat fraction | 30 minutes
  Change in fat fraction (in %) in leg muscles from baseline to 6-year follow-up
Change in fibrosis in the heart | 1 hour
  Change in fibrosis (in %) in the heart from baseline to 6-year follow-up
Change in LVEF/GLS-score | 1 hour
  Change in LVEF/GLS-score (in %) in the heart from baseline to 6-year follow-up
Correlation between XCI and phenotype | 1 hour
  Correlation between XCI (ratio of healthy vs mutant X chromosome) and phenotype (from fat fraction and clinical symptoms). Correlation measured using linear regression.
Cardiac status in patients with BMD vs carriers of variants in the DMD gene | 1 hour
  Correlation between cardiac structure and function (measured through Dixon and spectroscopy from cardiac MRI) between patients with BMD and carriers of genetic variants of the DMD gene.

SECONDARY OUTCOMES:
Change in contractility | 1 hour
  Change in contractility (measured as the peak torque divided by the contractile cross sectional area of the muscle) in leg muscles from baseline to 6-year follow-up
Change in blood concentrations | 1 hour
  Change in blood concentrations of myoglobin(ng/ML)
Change in blood concentrations | 1 hour
  Change in blood concentrations of Creatine kinase(U/L)
Change in blood concentrations | 1 hour
  Change in blood concentrations of Creatine kinase MB(U/L)
Change in blood concentrations | 1 hour
  Change in blood concentrations of troponin T (TnT) (ng/ML)
Change in blood concentrations | 1 hour
  Change in blood concentrations of pro-brain natriuretic peptide (proBNP)(pg/ML)
Change in lower extremity strength | 1 hour
  Change in lower extremity strength(measured by biodex 4 in Nm) from baseline to 6-year follow-up.
Change in questionnaires on fatigue | 5 minutes
  Change in questionnaires on fatigue (using the fatigue severity scale score) from baseline to 6-year follow-up.
Progression of electrocardiographic findings | 10 minutes
  Progression of electrocardiographic findings from baseline to 6 year follow-up (measured by electrocardiographic as number of new incidents)
Correlation between cardiac structure and function | 1 hour
  Correlation between cardiac structure (Dixon and spectroscopy from cardiac MRI) and muscle function (measured through the medical research council score from 1-5) in patients with BMD

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen neuromuscular center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No